CLINICAL TRIAL: NCT01718054
Title: Development of a Ready-to-use Nutraceutical Food for Patients With Sickle Cell Disease (SCD): Testing of Vascular Support Components
Brief Title: Vascular Function Intervention Trial in Sickle Cell Disease
Acronym: V-FIT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VFIT001; WT094780 (Other Grant/Funding Number: The Wellcome Trust, UK)
Record Dates: First submitted 2012-02-01; First posted 2012-10-31 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease
Keywords: Vascular function; Ready to use supplementary foods; Chloroquine; Children; Growth; Nitric Oxide
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vascular (Active Comparator): In this intervention period children will receive a vascular ready-to-use supplementary food with added L-Arginine & L-Citrulline plus daily chloroquine
  Interventions: Dietary Supplement: Vascular ready-to-use supplementary food; Drug: Chloroquine
- regular (Active Comparator): In this intervention period children will receive a regular ready-to-use supplementary food plus weekly dose of chloroquine
  Interventions: Dietary Supplement: Regular Ready-to-use supplementary food; Drug: Chloroquine

INTERVENTIONS:
Dietary Supplement: Vascular ready-to-use supplementary food — Daily vascular ready-to-use supplementary food containing protein, energy and fortified with 1 x recommended daily allowance(RDA) of vitamins and minerals except for folic acid = 1mg and with no iron fortificant included and fortified with arginine and citrulline amino acids
  Arms: vascular
Dietary Supplement: Regular Ready-to-use supplementary food — Daily ready-to-use supplementary food containing protein, energy and fortified with 1 x RDA vitamins and minerals except for folic acid = 1mg and with no iron fortificant included.
  Arms: regular
Drug: Chloroquine
  Other Names: Malaviron syrup

SUMMARY:
Sickle cell disease (SCD) is the most common inherited disorder worldwide affecting 300,000 births annually, most occuring in sub-Saharan Africa (SSA) where poor detection and care result in high childhood mortality, malnutrition, illness and disability in survivors. SCD is caused by abnormal haemoglobin, the compound in red blood cells(RBC) that carries oxygen. Much of the disability in SCD may be caused by vascular damage from the breakdown of damaged RBC. Research in high-income countries has led to some effective therapies but these are currently costly and complex. The investigators will test two different formulations of an affordable, ready-to-use supplementary food (RUSF) specifically tailored for children with SCD. As well as containing energy, protein, essential fats, vitamins and minerals, the vascular RUSF (RUSFv) will be fortified with the amino-acids arginine and citrulline and be delivered with a daily chloroquine dose to create a novel "nutraceutical" intervention. Arginine is converted to nitric oxide which is essential for vascular health. Arginine levels are low in SCD because the arginine-degrading enzyme, arginase, is released from RBCs. The investigators propose that by supplying additional arginine (and citrulline which converts to arginine) and suppressing arginase activity (an action of chloroquine) the investigators can improve vascular function. Our study will test this theory, and if provision of RUSF improves growth in children with SCD.

DETAILED DESCRIPTION:
Arginine is the substrate of endothelial nitric oxide (NO) synthase. Citrulline converts to arginine and has a greater bioavailability than arginine. Chloroquine is a competitive inhibitor of arginase which is released from lysed red cells and possibly through liver damage. Raised arginase predicts low plasma arginine levels and may predict clinical disease severity.

The interventions being tested are designed to target:

(i) the moderate to severe growth retardation commonly observed in children with SCD especially in low income countries; (ii) endothelial dysregulation secondary to low NO bioavailability, inflammation and oxidant stress, hypothesised to underlie much of the clinical pathology in SCD.

This study will test the following hypotheses:

1. That the provision of energy, protein and micronutrients within a ready to use supplementary food will increase linear growth, weight gain and proportion of fat-free mass in children with SCD.
2. That the provision of supplementary L-arginine and L-citrulline within the matrix of a twice-daily RUSF plus daily chloroquine (CQ) for 4 months, compared to a standard RUSF and weekly anti-malarial prophylaxis CQ to children with SCD will:

   * Increase plasma arginine concentrations and the ratio of plasma arginine: ornithine.
   * Decrease or not alter plasma asymmetric dimethylarginine (ADMA) concentrations
   * Improve NO-dependent vascular function as detected by an increase in maximum flow mediated dilatation (FMDmax)
3. That the provision of daily CQ at a dosage of 2-3mg base/kg/day for 4 months to children with SCD will:

   * Decrease the activity of plasma arginase through competitive inhibition
   * Decrease levels of plasma inflammatory markers

If successful then larger studies of efficacy and effectiveness would be needed to assess long-term endpoints of hospitalization, stroke, and mortality. Existing evidence suggests that the proposed intervention also has the potential to increase the efficacy of hydroxyurea (HU) therapy. The successful development of an affordable ready-to-use 'nutraceutical' food with proven efficacy in growth promotion and vascular health could represent a major step forward for SCD patients in low-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-11 years old at enrolment and resident within urban Dar-es-Salaam
* Enrolled in Muhimbili Sickle Cohort and attending routine Muhimbili National Hospital sickle clinics
* Homozygous for hemoglobin S (HbSS) phenotype confirmed by electrophoresis and high performance liquid chromatography (HPLC)

Exclusion Criteria:

* >95th percentile for body mass index (BMI) for age using British 1990 growth standards
* Receiving hydroxyurea therapy or significant other long-term drug therapy
* Diagnosis with clinically significant non-SCD related disease including:

  * Stage III or above HIV - or receiving ART therapy regardless of AIDS stage
  * Tuberculosis infection
* Blood transfusion within previous 30 days
* Previously diagnosed clinical pulmonary hypertension or cardiac dysfunction or clinical signs of pulmonary hypertension (loud pulmonary second heart sound) or heart failure (displaced apex beat, high jugular venous pressure, enlarged liver, peripheral oedema)
* Low visual acuity at baseline (<6/9 using a modified (for Tanzania) Snellen chart or previously diagnosed chronic eye disorder likely to suggest retinopathy or macular degeneration
* Significant hepatic/renal dysfunction assessed by clinical chemistry panel at baseline
* Epilepsy, psoriasis or currently taking any drugs listed as interacting with chloroquine

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
ratio of arginine to ornithine concentration & ratio of arginine to ADMA | 4 or 12 months
  We will compare the effects of the RUSFv compared to the simple RUSF on:
  The ratio of plasma arginine to ornithine & ratio of arginine to ADMA and adjust for values at baseline
  Time frame definition:
  0 months = baseline
  4 months = after 1st four-month intervention period, before washout 1
  8 months = after 1st 4 month washout period before 2nd intervention period
  12 months = after 2nd four-month intervention period, before washout 2
  16 months = after 2nd 4 month washout period (study end)
Nitric Oxide dependent endothelial function | months 4 or 12
  Comparison of the effects of the RUSFv to the simple RUSF on vascular function, assessed using flow mediated dilatation (FMDmax), adjusted for baseline values at time 0. Values will also be determined at time point at month 8, in order to check for possible carry-over effect.
Linear Growth and Weight Gain | After 8 months of treatment with RUSFv and RUSF
  We will compare the effects of RUSF compared to no RUSF on rates of growth by comparison of the 2 intervention periods combined with the two washout periods combined, by conducting measurements at months 0, 4, 8, 12 & 16.

SECONDARY OUTCOMES:
Haemoglobin concentration | months 0, 4, 8, 12 & 16
  Full blood counts (FBC) of ethylenediaminetetraacetic acid (EDTA) whole blood will be conducted
Markers of inflammation and vascular activation | months 0, 4 & 12
  Concentrations of soluble adhesion molecules (VCAM-1, vascular endothelial growth factor-1 (VEGF-1), tumor necrosis factor-alpha (TNF-α) & e-selectin, tissue factor and IL-6) will be measured in frozen (-80⁰C) plasma aliquots.
  C-reactive protein concentrations will be measured in frozen serum samples and leukocyte counts from FBC.
Markers of haemolysis | months 0, 4 & 12
  Plasma haemoglobin will be measured in frozen serum aliquots. Unconjugated bilirubin and lactate dehydrogenase in fresh serum.
Frequency of vaso-occlusive painful episodes | Weekly from month 0-16
  Study personnel will administer detailed questionnaires at weekly home visits to assess the frequency of all sickle and non-sickle associated morbidity and health seeking behaviour, with a focus on painful episodes. Participatory research will be used to determine the likely application and optimal formatting of pain diaries to be completed by patients and families in addition to the standard questionnaire.
liver and kidney function clinical chemistry | months 0, 4 & 12
  aspartate transaminase, alkaline phosphatase, total and direct bilirubin and creatinine will be measured in fresh serum
glomerular filtration rate | months 0, 4 and 12
  glomerular filtration rate will be estimated using an adaptation of the Schwartz equation in which muscle mass measured using bioimpedance will be included in the formula instead of the usual estimate. The outcome will be adjusted for values at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cox, PhD, Principal Investigator — London School of Hygiene & Tropical Medicine, UK / Muhimbili Wellcome Programme, Tanzania
Locations (1):
- Muhimbili University of Heath and Allied Sciences (MUHAS), Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Cox SE, Ellins EA, Marealle AI, Newton CR, Soka D, Sasi P, Luca Di Tanna G, Johnson W, Makani J, Prentice AM, Halcox JP, Kirkham FJ. Ready-to-use food supplement, with or without arginine and citrulline, with daily chloroquine in Tanzanian children with sickle-cell disease: a double-blind, random order crossover trial. Lancet Haematol. 2018 Apr;5(4):e147-e160. doi: 10.1016/S2352-3026(18)30020-6. Epub 2018 Mar 13. PMID 29548623